CLINICAL TRIAL: NCT05406063
Title: Stereotactic Multiple Fraction Radiotherapy for Non-spine Bone Metastases a Multicentre Prospective, Open Label, Randomised Controlled Phase 3 Non-inferiority Clinical Trial
Brief Title: Stereotactic Multiple Fraction Radiotherapy for Non-spine Bone Metastases
Acronym: SMILE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Collaborators: Krebsforschung Schweiz, Bern, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00631
Record Dates: First submitted 2022-05-03; First posted 2022-06-06 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Radiation Therapy; Bone Metastases; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT with 9 Gy x 3 fractions to the treatment site. (Experimental): Patients will be treated with SBRT delivering 9 Gy x 3 fractions (BED10: 51.3 Gy) to the treatment site.
  Interventions: Radiation: SBRT
- SBRT with 7 Gy x 5 fractions to the treatment site (Active Comparator): Patients will be treated with SBRT delivering 7 Gy x 5 fractions (BED10: 59.5 Gy) to the treatment site.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Stereotactic multiple fraction radiotherapy

SUMMARY:
To investigate, whether multi-fraction stereotactic body radiation therapy (SBRT) within 3 treatment fractions is non-inferior to the current standard of care of 5 fraction SBRT regarding pain response at 3 months after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Personally signed and dated written informed consent,
* Histological diagnosis of malignancy,
* Histologically or radiologically diagnosed bone metastasis,
* Age ≥ 18 years
* Pain or under pain control medication

Exclusion Criteria:

* Pregnant or lactating women,
* Women of childbearing potential or sexually active males not willing to use effective contraception while on treatment and 3 months after the end of treatment,
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc.,
* Prior radiotherapy to the intended treatment site,
* Lesions > 5cm in maximum diameter,
* Prior treatment with radioactive isotopes within 30 days of randomisation,
* Spinal column, hands, feet, or head as intended treatment site,- Fracture at the intended treatment site,
* Surgery required or previous surgery at the intended treatment site
* Instability of the intended treatment site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain relief (response rate) measured with the Visual Analog Scale (VAS) from Baseline to 3 months after treatment. | Baseline and 3 months after treatment
  The Visual Analog Scale is a validated, subjective measure for pain. Possible scores ranges between zero (no pain) and ten (worst possible pain).
  The primary endpoint was defined as pain relief > 2 points from Baseline to 3 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Foerster, MD, Principal Investigator — Kantonsspital Winterthur KSW
Locations (2):
- Switzerland (2):
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - University Hospital Bern, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foerster R, Zwahlen DR, Schroeder C, Windisch P, Halatsch ME, Alfieri A, Meier C, Hemmatazad H, Aebersold DM, Buchali A, Habermehl D, Batifi N. SMILE-stereotactic multiple fraction radiotherapy for non-spine bone metastases: study protocol for a multicenter, open-label phase III randomized controlled trial. Trials. 2024 Nov 13;25(1):762. doi: 10.1186/s13063-024-08608-6. PMID 39538259